CLINICAL TRIAL: NCT00769808
Title: A Prospective Trial to Evaluate the Safety and Effectiveness of the Bausch & Lomb Technolas® 217z Laser With Zyoptix® Aspheric Algorithm When Used for the LASIK Treatment of Myopia and Myopic Astigmatism
Brief Title: Technolas 217z Laser With Zyoptix Aspheric Algorithm Used for the LASIK Treatment of Myopia and Myopic Astigmatism.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 564
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-08

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: This was a medical device study with only one intervention used for lasik correction surgery
Oversight: Data Monitoring Committee: No

ARMS (1):
- Technolas 217z Excimer Laser (Experimental): Bausch & Lomb Zyoptix Aspheric Algorithm for LASIK correction of myopia and myopic astigmatism.
  Interventions: Device: Bausch & Lomb 217z Excimer Laser

INTERVENTIONS:
Device: Bausch & Lomb 217z Excimer Laser — LASIK correction of myopia and myopic astigmatism

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Bausch & Lomb Technolas 217z laser with the investigational Zyoptix Aspheric Algorithm when used for LASIK treatment of myopia and myopic astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were of legal age (at least 18) and had full legal capacity to volunteer.
* Subjects must be willing to have both eyes treated with the laser.
* Subjects must have up to -12.00D of absolute spherical myopia (not spherical equivalent) with up to -6.00D of refractive astigmatism, with a spherical equivalent up to -15.00D as measured by manifest subjective refraction.
* Subjects who had less than 0.75 D of difference in the preoperative manifest spherical equivalent and cycloplegic spherical equivalent subjective refractions.

(Manifest subjective refractions adjusted for optical infinity were used.)

* High contrast, manifest best spectacle-corrected distance logMAR visual acuity correctable to at least 0.3 in both eyes, and must not differ between eyes by more than 1 line (5 letters).
* Contact lens wearers must have 2 Orbscan measurements and 2 manifest subjective refractions taken preoperatively at least 1 week apart.
* Contact lens wearers must have gas permeable lenses discontinued for at least 3 weeks and soft lenses discontinued for at least 2 weeks prior to the preoperative evaluation.

Exclusion

* Subjects with uncorrected visual acuity better than 20/40 (Snellen) or 0.3 logMAR
* Subjects who were immuno-compromised or had a diagnosis of connective tissue disease, clinically significant atopic disease, diabetes, autoimmune diseases and other acute or chronic illnesses that increased the risk to the subject or could have confounded the outcomes of this study.
* Subjects with uncontrolled glaucoma or glaucoma who were under treatment in the study eye or with ocular hypertension.
* Subjects who demonstrated evidence of retinal vascular disease.
* Subjects who have an ocular muscle disorder including strabismus or nystagmus, or other disorders that affected fixation.
* Subjects who were at risk for angle closure or who had a potentially occludable angle, as evidenced by a shallow anterior chamber on slit lamp exam, confirmed by gonioscopy as deemed necessary by the study Investigator.
* Subjects who had undergone previous intraocular or corneal surgery of any kind, including any type of excimer laser surgery for either refractive or therapeutic purposes.
* Subjects who were taking systemic medications likely to affect wound healing such as corticosteroids or anti-metabolites or any other medications that may increase the risk to the subject or confound the outcomes of this study.
* Subjects for whom the combination of their preoperative corneal thickness and the planned operative parameters for the LASIK procedure could have resulted in less than 250 microns of remaining posterior corneal thickness below the flap postoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cohen, MD, Principal Investigator — Lasik MD
Locations (1):
- Lasik MD, 130 King Street, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy two myopic participants (144 eyes) were enrolled.
Period: Overall Study
Arm/Group | Technolas 217z Excimer Laser
Started | 72
Completed | 64
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: Participants receiving treatment and demographic data.
Arm/Group | Technolas 217z Excimer Laser
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 40
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Uncorrected High Contrast Distance Visual Acuity of 20/40 or Better
Time Frame: 3 months
Population: There were 59 participants with visual acuity data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Excimer Laser
Number analyzed (Participants) | 59
Number analyzed (eyes) | 118
percentage of eyes | 99.2 [97.5 to 100]

2. Primary Outcome: Percentage of Eyes With Manifest Subjective Refraction (MRSE) Within ± 1.00 Diopter (D) and 0.50 D of Emmetropia
Description: Manifest refractions (eyeglass prescriptions) have three components: sphere, cylinder, and axis. Sphere and cylinder are both expressed in diopters, which is a continuous measure of the focusing power needed to make the image sharp on the retina. Manifest refraction spherical equivalent (MRSE) is equal to sphere + ½ x cylinder. It is expressed in diopters (D).
Time Frame: 3 months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Excimer Laser
Number analyzed (Participants) | 59
Number analyzed (eyes) | 118
eyes
  Within 0.50 D | 109
  Within 1.00 D | 117

3. Primary Outcome: Preservation of Manifest Best Corrected High Contrast Distance Visual Acuity
Description: Mean change in best-corrected high contrast distance visual acuity. Corrected means spectacle corrected. Visual acuity (VA) was reported as letters read correctly, and the letters read were converted to logarithm of the minimum angle of resolution (logMAR) acuity. The participant read rows of letters on a standard LogMAR chart until the participant misses 3 letters on a row with 5 letters. The total number of correct letters were recorded. A decrease in the number of correct letters indicates a decrease in visual acuity. Acuity was averaged across visits.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Excimer Laser
Number analyzed (Participants) | 59
Number analyzed (eyes) | 118
units on a scale | -0.055 (0.103)

4. Primary Outcome: Percentage of Eyes With Manifest Best-corrected Distance Photopic Visual Acuity Decrease of 2 or More Lines
Time Frame: 3 months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Excimer Laser
Number analyzed (Participants) | 59
Number analyzed (eyes) | 118
eyes | 1

5. Primary Outcome: Percentage of Eyes With > 2.00 Diopter of Induced Postoperative Refractive Cylinder
Description: as for outcome 2
Time Frame: 3 months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Excimer Laser
Number analyzed (Participants) | 59
Number analyzed (eyes) | 118
eyes | 0

6. Primary Outcome: Percentage of Eyes That Had High Contrast Best Spectacle Corrected Visual Acuity (HCBSCVA) of 20/20 or Better at Baseline Had a Visual Outcome Worse Than 20/40 at 3 Months
Description: Corrected means spectacle corrected. Visual acuity (VA) was reported as letters read correctly, and the letters read were converted to logarithm of the minimum angle of resolution (logMAR) acuity. The participant read rows of letters on a standard LogMAR chart until the participant misses 3 letters on a row with 5 letters. The total number of correct letters were recorded. A decrease in the number of correct letters indicates a decrease in visual acuity. Acuity was averaged across visits.
Time Frame: 3 months
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Excimer Laser
Number analyzed (Participants) | 59
Number analyzed (eyes) | 118
eyes | 0

7. Secondary Outcome: Percentage Change From Baseline in Higher Order Aberrations.
Description: The aberrations in the eye's optical system were measured over the entire pupil by the Bausch & Lomb Zywave II WaveFront Aberrometer, a Hartmann-Shack type device. The pupil should have been at least 6 mm in diameter using 2.5% phenylephrine as a dilating agent to maximize the pupil diameter and hence the amount of wavefront information collected by the Zywave II. The wavefront data was then fitted with Zernike polynomials representing the 2nd, 3rd, 4th and 5th order Zernike terms. These terms represent the wavefront aberration of the eye.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: Percentage change
Units Other Than Participants: eyes
Arm/Group | Technolas 217z Excimer Laser
Number analyzed (Participants) | 59
Number analyzed (eyes) | 118
Percentage change | 24.9 (0.1413)

ADVERSE EVENTS:
Time Frame: 6 months
Description: There were 66 treated participants evaluated for adverse events.
Arm/Group | Technolas 217z Excimer Laser
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 51/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Technolas 217z Excimer Laser (N=66)
Bowman's membrane disorder (Eye disorders) | 8
Corneal edema (Eye disorders) | 4
Keratitis (Eye disorders) | 16
Punctate keratitis (Eye disorders) | 36
Eye operation complication (Eye disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other